CLINICAL TRIAL: NCT01580982
Title: Molecular Analysis of Oncogenes and Resistance Mechanisms in Lung and Other Thoracic Cancers
Brief Title: Molecular Analysis of Oncogenes and Resistance Mechanisms in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-1621.cc
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasms
Keywords: Oncogenes; Lung and Other Thoracic Cancers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue will be acquired from either archival or de novo biopsy material
Oversight: Data Monitoring Committee: No

SUMMARY:
The mechanisms of sensitivity and resistance to oncogene-targeted therapy can be determined from tumor tissue or tumor cell lines derived from available archival samples and/or from standard-of-care re-biopsy upon suspected tumor progression.

DETAILED DESCRIPTION:
To identify baseline and treatment-related somatic changes in the tumor tissue from patients with lung and other thoracic cancers. To estimate the proportion of patients that subsequent therapy is altered based on the information acquired from such biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing investigation or treatment for thoracic cancers with oncogene-targeted therapies
2. Aged 18 years or older
3. Either a) have suspected tumor progression or other condition that dictates a standard-of-care palliative, therapeutic, or diagnostic intervention including but not limited to procedures such as bronchoscopic biopsy, computed tomography (CT) or ultra-sound (US)-guided biopsy, thoracentesis, video assisted thoracoscopic (VATS) pleurodesis, lobectomy, adrenalectomy or pleural catheter placement, providing tumor specimen appropriate molecular analysis or b) have previously had biopsy/surgical intervention with tumor tissue at University of Colorado or an outside institution available for medullar analysis.
4. Patients must have the ability to understand and willingness to sign an informed consent document.

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered for this study would be undergoing a standard care procedure
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01-23 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To identify baseline and treatment-related somatic changes in the tumor tissue from patients with lung and other thoracic cancers. | To be determined upon funding

SECONDARY OUTCOMES:
To estimate the proportion of patients that subsequent therapy is altered based on the information acquired from such biopsies | To be determined upon funding

CONTACTS AND LOCATIONS:
Overall Officials: Erin Schenk, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided